CLINICAL TRIAL: NCT00685529
Title: An Open-Label, Randomized, Multiple Dose, 3-Way Crossover Study of Arformoterol Tartrate Inhalation Solution and Foradil® (Racemic Formoterol) in Subjects With Mild to Moderate Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Study of Arformoterol Tartrate Inhalation Solution and Racemic Formoterol in Subjects With Mild to Moderate Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 091-019
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: COPD
Keywords: COPD; Arformoterol; formoterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): 12 µg of racemic formoterol fumarate BID
  Interventions: Drug: Racemic formoterol
- B (Experimental): 15 µg of nebulized arformoterol tartrate inhalation solution BID
  Interventions: Drug: Arformoterol tartrate inhalation solution
- C (Active Comparator): 24 µg of racemic formoterol fumarate BID
  Interventions: Drug: Racemic formoterol

INTERVENTIONS:
Drug: Racemic formoterol — 12 µg of racemic formoterol fumarate BID
  Other Names: Foradil®; Aerolizer
  Arms: A
Drug: Arformoterol tartrate inhalation solution — 15 µg of nebulized arformoterol tartrate inhalation solution BID
  Other Names: Brovana, (R,R)-formoterol
  Arms: B
Drug: Racemic formoterol — 24 µg of racemic formoterol fumarate BID
  Other Names: Foradil®; Aerolizer
  Arms: C

SUMMARY:
The purpose of this study is to compare the blood levels of arformoterol tartrate inhalation solution to racemic formoterol in male and female subjects with mild to moderate Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
This is an open label, randomized, multiple dose, 3-way crossover, multicenter, inpatient and outpatient study to compare the pharmacokinetic (PK) profile of arformoterol tartrate inhalation solution and Foradil® in male and female subjects with mild to moderate COPD. Up to 36 subjects (with a minimum 40% of each gender) were to be randomized to ensure that at minimum 24 subjects completed the study. The study included 3 dose periods and 3 washout periods. Subjects received 3 different treatments in random order for 13 consecutive days and a single dose on the morning of the 14th day. Subjects will be randomly assigned to 1 of the 6 possible treatment sequences. During each dose period, subjects received medication via nebulization or DPI twice daily for 13 consecutive days and a single dose on the morning of the 14th day. There was be a 10 day washout period between each treatment. Subject participation was be approximately 13 weeks and included a screening visit and 7 study visits. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects must be at least 35 years old at the time of consent.
* Female subjects less than or equal to 65 years old must have a negative serum pregnancy test at Visit 1 and a urine pregnancy test at Visit 2, confirmed negative prior to randomization. Subjects of childbearing potential must be using an acceptable method of birth control.
* Subjects must have a documented primary clinical diagnosis of non-asthmatic COPD
* Subjects must have a ≥ 15 pack-year smoking history
* Subjects must be in general good health.
* Subjects must have a minimum blood pressure of 105/60 mmHg and a minimum resting pulse of 50 bpm at Screening Visit 1.
* Subjects must have a body mass index (BMI) of at least 16 kg/m2 but no more than 30 kg/m2. (BMI is defined as the subject's weight in kilograms divided by the square of the subject's height in meters.)
* Subjects must be willing to remain in the residential facility for 3 separate 24 hour visits and 3 separate 36-hour visits.
* Subjects must agree to refrain from strenuous activities, as defined by the Principal Investigator, throughout the study, from the screening visit until after the end of study/early termination visit.

Exclusion Criteria:

* Subject has had a febrile illness within 72 hours (3 days) before Screening.
* Subject has any clinically significant unstable medical abnormality, chronic disease, or a history of a clinically significant abnormality of the cardiovascular, respiratory, gastrointestinal, hepatic, or renal systems, which, in the opinion of the investigator, may affect the safety of the subject.
* Subject has a history of malignancy or currently has malignancy other than non melanomatous skin cancer. Subjects who have been cancer-free for 5 years or more may be enrolled.
* Subjects with a chest x-ray that suggests a diagnosis other than COPD (e.g., diagnostic of pneumonia, other infection, atelectasis, or pneumothorax or other active/ongoing pulmonary conditions) and taken within 6 months prior to study start. If there is no chest x-ray taken within 6 months prior to study start, or if recent results are unavailable for review, a chest x-ray must be performed.
* Subjects with a history of asthma, with the exception of asthma diagnosed in childhood.
* Subject tests positive at screening for hepatitis B surface antigen or hepatitis C antibody, or the subject has a history of a positive result.
* Subject is known to be seropositive for human immunodeficiency virus (HIV).
* Female subject is pregnant or lactating.
* Female subject who (a) is of childbearing potential and not using contraception or is using hormonal contraception, or (b) is post-menopausal and is taking any form of hormone replacement therapy.
* Subject has a disorder or history of a condition that may interfere with drug absorption, distribution, metabolism, or excretion (e.g., malabsorption, gastrointestinal surgery).
* Subject has participated in any investigational study within 30 days prior to screening or is currently participating in another clinical trial.
* Subject is a staff member or relative of a staff member.
* Subject has a positive urine alcohol test during screening. Subjects with a known history of alcohol use may be enrolled in the study if the subject's alcohol use is not indicative of abuse. Abuse is defined as current consumption of more than three alcoholic beverages per day.
* Subject has a history or suspected history of abuse of a barbiturate, amphetamine, or narcotic and/or has a positive screening result for any of these substances at study start.
* Subject has a history of allergic reaction to the study medication or any components of the study medications.
* Subject has received oral anticoagulant therapy within 90 days before Screening.
* Subject has had significant blood loss (>500 cc) or donated blood within 60 days preceding screening or plans to donate blood during or within 60 days after completing the study.
* Subject has donated plasma within 72 hours prior to the first dose of study drug.
* Subject has had an acute illness within 10 days of Day 1.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-04; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for this study is exposure to (R,R)-formoterol, measured by the PK parameters AUC(0-τ) and Cmax | Treatment/Washout 1: Days 1, 12-18; T/W 2: 24, 35-40; T/W 3: 47, 58-64, EOT: 70

SECONDARY OUTCOMES:
Additional PK parameters of (R,R)-formoterol include tmax, t ½, and AUC(0-∞) | Treatment/Washout 1: Days 1, 12-18; T/W 2: 24, 35-40; T/W 3: 47, 58-64, EOT: 70
Accumulation ratios for (R,R)-formoterol as measured by RCmax and RAUC(0-τ) | Treatment/Washout 1: Days 1, 12-18; T/W 2: 24, 35-40; T/W 3: 47, 58-64, EOT: 70
PK parameters for (S,S)-formoterol following racemic formoterol administration are AUC(0-τ), Cmax, tmax, t ½, and AUC(0-∞) | Treatment/Washout 1: Days 1, 12-18; T/W 2: 24, 35-40; T/W 3: 47, 58-64, EOT: 70
Accumulation ratios for (S,S)-formoterol as measured by RCmax and RAUC(0-τ) | Days 1, 12, 13, 14, 15, 16, 17,18
FEV1 and % predicted FEV1 | Treatment/Washout 1: Days 1, 14-15; TW2: 24, 37-38; TW3: 47, 60-61

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Long Beach, California
  - Fort Lauderdale, Florida
  - Raleigh, North Carolina
  - Simpsonville, South Carolina
  - Spartanburg, South Carolina
  - Spokane, Washington